CLINICAL TRIAL: NCT02460770
Title: Pilot Study of Investigation of Bone Marrow-derived Mesenchymal Stem Cells (MSC) Administration in Weaning From Left Ventricular Assist Device
Brief Title: Bone Marrow-derived Mesenchymal Stem Cells (MSC) Administration in Weaning From Left Ventricular Assist Device
Acronym: MESAD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Thoratec Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13 150 03
Record Dates: First submitted 2015-01-22; First posted 2015-06-02 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Chronic Myocardial Ischemia
Keywords: Left Ventricular Assist Device; stem cell therapy; ischemic heart failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous mesenchymal stem cells (Experimental): After bone-marrow aspiration by an authorized person, Mesenchymal Stem Cells were isolated and cultured during 17 days by the French Blood Establishment. Then, patients receive intramyocardial injections of Mesenchymal Stem Cells during Left Ventricular Assist Device surgery
  Interventions: Drug: Autologous mesenchymal stem cells

INTERVENTIONS:
Drug: Autologous mesenchymal stem cells — After bone-marrow aspiration by an authorized person, mesenchymal stem cells were isolated and cultured during 17 days by the French Blood Establishment. Then, patients receive intramyocardial injections of mesenchymal stem cells during device surgery.
  Other Names: MSC

SUMMARY:
Left Ventricular Assist Devices are commonly used to assist failing hearts as a bridge to transplantation or for long-term support. The purpose of the MESenchymal stem cell therapy and Left Ventricular Assist Device program is to improve heart function with stem cell therapy and attempt to wean patients from HeartMate Left Ventricular Assist Device.

DETAILED DESCRIPTION:
Currently Left Ventricular Assist Device-only patients are being implanted and followed. Feasibility of autologous mesenchymal stem cell grafting in patients receiving heart mate will be assessed in a 4 patient pilot trial. Mesenchymal stem cell are delivered during Left Ventricular Assist Device surgery by intramyocardial infusions. Recovery of contractile function of the heart is assessed during attempts to wean patients from Left Ventricular Assist Device

ELIGIBILITY:
INCLUSION CRITERIA:

* Postmenopausal female or female who may become pregnant but is using adequate contraceptive precautions with negative pregnancy test,
* Severe Left Ventricular dysfunction with Ejection Fraction < 30% with ischemic cardiomyopathy,
* New York Heart Association Class III or IV,
* No revascularization options available,
* Listed or not for cardiac transplantation,
* Clinical indication and accepted candidate for Left Ventricular Assistance Device implantation as a destination therapy or as a bridge to transplantation,
* Optimal medical therapy.

EXCLUSION CRITERIA:

* Cardiothoracic surgery within 30 days prior to study entry,
* Myocardial infarction within 3 months prior to study entry,
* Prior cardiac transplantation,
* Left Ventricular reduction surgery or cardiomyoplasty,
* Acute reversible cause of heart failure (e.g. myocarditis, profound hypothyroidism),
* Left ventricular aneurysm or wall thickness preventing cell injections,
* Anticipated requirement for biventricular mechanical support,
* Stroke within 30 days prior to study entry,
* Received investigational intervention within 30 days of study entry,
* Pregnant or breastfeeding at time of study entry,
* Human Imune deficiency Virus, Human T-cell Lymphotrophic Virus, Hepatitis B Virus and Hepatitis C Virus positive within 30 days prior to study entry,
* Active systemic infection within 48 hours prior to study entry,
* History of cancer in the last 5 years,
* Patient participant to other research,
* Patient under treatment that may exert an inhibitory or stimulatory effect on the growth and multiplication of cells, or with immunosuppressive properties.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Estimated); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of the full procedure | 1 month
  ability to perform bone marrow aspiration, cell culture and intramyocardial injections during left Ventricular Assist Device surgery Realization of a full injection procedure

SECONDARY OUTCOMES:
Ejection Fraction | 12 months
  Global and regional contractile function during echocardiography
Maximal Oxygen consumption | 12 months
  Maximum rate of oxygen consumption as measured during incremental exercise, modification of the body mass (muscular lean mass, muscular strength), duration of the test and load,
Walking distance in 6 minutes | 12 months
  measure of walk distance during six minutes
weaning procedure | 12 months
  progressive reduction of the pump speed
Quality of life | 12 months
  assessment of quality of life by Minnesota Living with Heart Failure Questionnaire
Measure of heart pressures | 12 months
  measure of heart pressures and cardiac output
Brain natriuretic peptide | 12 months
  assessment of variation of brain natriuretic peptide
Troponin | 12 months
  assessment of variation of troponin
Major bleeding | 1 month
Systemic embolism | 1 month
Deaths | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Roncalli Jérome, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Cardiology Department of Rangueil Hospital - Rangueil Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided